CLINICAL TRIAL: NCT07334093
Title: A Multicenter, Randomized Controlled Phase II Clinical Study of Hetrombopag Combined With rhTPO in the Treatment of Cancer Therapy-induced Thrombocytopenia (CTIT) in Solid Tumor Patients.
Brief Title: A Study of Hetrombopag Combined With rhTPO in the Treatment of Cancer Therapy-induced Thrombocytopenia (CTIT) in Solid Tumor Patients.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Yanxia, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2025-803-01
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Cancer Therapy-induced Thrombocytopenia (CTIT)
MeSH Terms: interventions — hetrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): rhTPO 15,000 IU/day subcutaneously + hetrombopag 7.5 mg/day orally, both starting on Day 1 for up to 14 days.
  Interventions: Drug: rhTPO + hetrombopag
- Control arm (Active Comparator): Hetrombopag 7.5 mg/day orally starting on Day 1 for up to 14 days.
  Interventions: Drug: hetrombopag

INTERVENTIONS:
Drug: rhTPO + hetrombopag — rhTPO 15,000 IU/day subcutaneously + hetrombopag 7.5 mg/day orally, both starting on Day 1 for up to 14 days.
  Arms: Experimental arm
Drug: hetrombopag — Hetrombopag 7.5 mg/day orally starting on Day 1 for up to 14 days.
  Arms: Control arm

SUMMARY:
Objective To evaluate the efficacy and safety of hetrombopag plus rhTPO versus hetrombopag monotherapy for CTIT in solid-tumor patients.

Participants 204 histologically- or cytologically-confirmed solid-tumor patients with ≥grade 3 thrombocytopenia following anti-cancer treatment.

Design

Open-label, multicenter, randomized controlled phase II study. Patients are randomized 1:1 into two arms:

Experimental arm (N=102):

rhTPO 15,000 IU/day subcutaneously + hetrombopag 7.5 mg/day orally, both starting on Day 1 for up to 14 days.

Control arm (N=102):

Hetrombopag 7.5 mg/day orally starting on Day 1 for up to 14 days. Stopping & Rescue Rules Stop study drug if PLT ≥100×10⁹/L or rises ≥50×10⁹/L from baseline. If PLT ≤10×10⁹/L or <20×10⁹/L with bleeding risk, give rescue therapy (platelet transfusion or investigator-chosen alternative).

Primary Endpoint Proportion of patients achieving PLT ≥100×10⁹/L or an increase ≥50×10⁹/L from baseline within 14 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years (inclusive), both sexes eligible.
2. Histologically or cytologically confirmed malignant solid tumor (e.g., lung, breast, gastric, colorectal, genitourinary cancers, etc.).
3. Currently receiving anti-cancer therapy: chemotherapy, radiotherapy, immuno-chemotherapy, targeted therapy, or combinations.
4. Grade ≥3 cancer-therapy-induced thrombocytopenia (PLT <50×10⁹/L).
5. ECOG performance status 0-1.
6. Estimated life expectancy ≥12 weeks.
7. Women of child-bearing potential must have a negative serum pregnancy test within 7 days before first dose and not be breastfeeding; they must agree to use effective contraception from enrollment through 7 days after the last study drug. Men with partners of child-bearing potential must be surgically sterilized or agree to use effective contraception during the same period and must not donate sperm.
8. Willing to participate, able to provide written informed consent, and expected to comply with the study protocol.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Individuals unable to understand the nature of the study or who have not given informed consent.
3. History of any arterial or venous thrombosis (stroke, transient ischemic attack, myocardial infarction, deep-vein thrombosis, pulmonary embolism) or clinical/laboratory evidence of a hypercoagulable disorder.
4. Cardiac disease within 3 months before screening: grade 3/4 congestive heart failure, arrhythmia requiring medication, myocardial infarction, conditions predisposing to thrombo-embolism (e.g., atrial fibrillation), or QTc prolongation.
5. Thrombocytopenia attributed to: concurrent chemoradiotherapy, non-anti-cancer therapy, oxaliplatin-induced sinusoidal injury, definite immune-mediated thrombocytopenia, severe bleeding symptoms, refractory persistent thrombocytopenia, or bone-marrow involvement proven by biopsy in patients with bone metastases.
6. Significant hepatic impairment:

   * No liver metastases: ALT/AST > 3 × ULN or TBL > 3 × ULN.
   * Liver metastases present: ALT/AST ≥ 5 × ULN or TBL ≥ 5 × ULN.
7. Known or anticipated hypersensitivity/intolerance to TPO-receptor agonists or any ingredient of hetrombopag ethanolamine tablets.
8. Concomitant use of other agents that may affect platelet count (e.g., traditional Chinese medicines, other thrombopoietic agents, antiplatelet drugs).
9. Receipt of any TPO-receptor agonist (eltrombopag, romiplostim, etc.), recombinant human TPO, or recombinant IL-11 within 1 month before screening.
10. Platelet transfusion within 3 days before randomization/first dose.
11. Any condition that, in the investigator's opinion, renders the patient unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-11-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving PLT ≥100×10⁹/L or an increase ≥50×10⁹/L from baseline within 14 days of treatment. | within 14 days of treatment.

SECONDARY OUTCOMES:
Proportion of patients achieving PLT ≥100×10⁹/L or an increase ≥50×10⁹/L from baseline within 7 days Time to PLT recovery to ≥100×10⁹/L Time to PLT increase ≥50×10⁹/L from baseline Lowest (nadir) platelet count recorded Duration of thrombopoietic therapy | within 7 days

IPD SHARING:
Plan to Share IPD: No